CLINICAL TRIAL: NCT01162915
Title: Phase I, Single Center, Trial to Asses Safety and Tolerability of the Intrathecal Infusion of Ex-vivo Expanded Bone-marrow Derived Mesenchymal Stem Cells for the Treatment of Spinal Cord Injury
Brief Title: Transfer of Bone Marrow Derived Stem Cells for the Treatment of Spinal Cord Injury
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Suspended due to lack of funding.
Sponsor: TCA Cellular Therapy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-SCI-I
Record Dates: First submitted 2010-07-13; First posted 2010-07-15 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2013-09

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Safety (Experimental): Infusion of autologous bone marrow-derived mesenchymal stem cells.
  Interventions: Biological: Autologous bone marrow-derived mesenchymal stem cells.

INTERVENTIONS:
Biological: Autologous bone marrow-derived mesenchymal stem cells. — Intrathecal infusion of a single dose of ex vivo expanded MSC.

SUMMARY:
This study is based on preclinical (animal) studies showing that infusing bone marrow-derived mesenchymal stem cells into the spinal fluid may contribute to improving neurologic function in animal models with spinal cord injuries. Bone marrow (BM) contains several types of stem cells that can produce functional cells. This includes cells that could help the healing process of damaged neurologic tissue.

The primary objective of this study is to see if the injection of these cells, obtained from your own bone marrow, is safe. A secondary objective is to evaluate if the treatment can provide functional improvements (neuromuscular control and sensation) in the affected areas.

DETAILED DESCRIPTION:
A Phase I, single-center trial to assess the safety and tolerability of an intrathecal infusion (lumbar puncture) of autologous, ex vivo expanded bone marrow-derived mesenchymal stem cells in a well-defined population of spinal cord injury patients.

Safety will be evaluated by neurological and non-neurological tests performed after short-term (1 to 30 days) and long-term (2 to 12 months)follow-up evaluation periods after cell infusion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65
* American Spinal Injury Association Impairment Scale A
* Clinical evidence of lesions located below c-spine 5 (C-5)
* Confirmation by MRI of injury level
* Time between injury and enrollment greater than 2 weeks
* Ability to provide informed consent
* Platelet count greater than 100 Thousand/uL at screening
* INR equal to or less than 1.5
* Hematocrit less than 30% prior to bone marrow aspiration
* Spinal cord injury within 60 months of screening

Exclusion Criteria:

* Anoxic brain injury
* Inability to provide consent
* Sepsis
* Neurological deficits attributed to lesions above C-5
* Cerebro-vascular accidents with intracranial hemorrhage, acute brain injuries, meningitis, hydrocephalus or other potential diseases where the pressure in the cerebro spinal fluid is increased
* Multiple sclerosis
* Amyotrophic lateral sclerosis
* Cerebral Palsy
* Evidence of cancer over the last 3 years prior to enrollment
* Immunosuppressive diseases
* Platelet count lower than 100,000
* White blood count greater than 15,000 unless the patient is on steroids
* Bleeding disorders
* Clinical or laboratory evidence of meningitis
* Skin infection at the infusion site
* Pregnant or planning to become pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-07; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Safety | 12 months
  Phase I trial to assess safety of intrathecal infusion of autologous mesenchymal stem cell treatment in spinal cord injury.

CONTACTS AND LOCATIONS:
Locations (1):
- TCA Cellular Therapy, LLC, Covington, Louisiana, United States

REFERENCES:
- See also: Related Info — http://www.tcacellulartherapy.com